CLINICAL TRIAL: NCT06660550
Title: Needlescopic Versus Traditional Laparoscopic Inguinal Hernia Repair in Pediatrics (A Prospective Comparative Study)
Brief Title: Needlescopic Versus Traditional Laparoscopic Inguinal Hernia Repair in Pediatrics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelaziz Ali Abdelaziz, M.B.B.Ch., Resident in Pediatric Surgery Department Sohag University Hospitals, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-15-10-4MS
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Congenital Inguinal Hernia

STUDY DESIGN:
Intervention Model Description: evaluate the results of Needlescopic inguinal hernia repair in comparison with traditional laparoscopic repair in children as regard operative time, cosmetic appearance, recurrence and other complications
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Needlescopic inguinal hernia repair (Active Comparator)
  Interventions: Procedure: Needlescopic inguinal hernia repair
- Traditional laparoscopic inguinal hernia repair (Active Comparator)
  Interventions: Procedure: laparoscopic inguinal hernia repair

INTERVENTIONS:
Procedure: laparoscopic inguinal hernia repair — traditional laparoscopic repair
  Arms: Traditional laparoscopic inguinal hernia repair
Procedure: Needlescopic inguinal hernia repair — Needlescopic inguinal hernia repair
  Arms: Needlescopic inguinal hernia repair

SUMMARY:
The aim of the study is to evaluate the results of Needlescopic inguinal hernia repair in comparison with traditional laparoscopic repair in children as regard operative time, cosmetic appearance, recurrence and other complications.

DETAILED DESCRIPTION:
Patients and methods:

* Place of the study: The study will be held in Department of Pediatric surgery in Sohag University Hospital.
* Type of the study: Prospective comparative Cohort study.
* Duration of the study: The study will last for 6 to 9 months starting from the date of acceptance of the protocol.
* Ethical considerations: The study will be carried out after approval by scientific and ethical committees of Sohag faculty of medicine.
* Method of the study:

Preoperative assessment:

1. Demographic data: e.g. name, age, sex …. etc.
2. History: e.g. complaint, present history and past surgical and medical history…etc.
3. General and local examination: e.g. laterality, associated anomalies …. etc.
4. Investigations:

Routine labs. Imaging: to confirm diagnosis in the affected side, to evaluate contralateral side, bilateral testicular volume as volumetric stander to evaluate testicular atrophy postoperative and other anomalies.

Operative technique:

Operative steps:

A. Traditional laparoscopic repair.

* STEPS:

  1. A 5mm port for the camera is introduced at umbilicus by open technique.
  2. Using triangulation rule to introduce two working ports.
  3. The abdomen is insufflated with carbon dioxide to 6-8 mmHg pressure in patients under 1 year of age and to 8-10 mmHg in older children.
  4. Diathermize the neck of the hernia sac with a diathermy hook.
  5. A 10-15 cm absorbable suture is passed into the peritoneal cavity through the abdominal wall next to the lateral port under vision.
  6. The purse-string stitch commences at the 2 o'clock position of the internal hernia opening.
  7. ensure that a "complete ring" of peritoneum has been included in the purse-string stitch without significant gaps.
  8. The purse-string suture is tied tightly using intracorporeally knot tying.

     B. Needlescopic Internal Ring Suturing.
* EQUIPMENT/SUTURE:

  1. One 5-mm trocar and 5-mm lens 30° or 0° telescope.
  2. Epidural needle.
  3. Non absorbable suture.
  4. Fascial closure instrument.
* STEPS:

  1. A 5mm port for the camera is introduced at umbilicus by open technique.
  2. The abdomen is insufflated with carbon dioxide to 6-8 mmHg pressure in patients under 1 year of age and to 8-10 mmHg in older children.
  3. The suture is introduced through the barrel of the epidural needle.
  4. Maintaining both ends of the preloaded suture extra peritoneal, the needle is advanced under the peritoneum around lateral half of the internal ring.
  5. The peritoneum is entered and the suture advanced into the abdominal cavity, creating a loop.
  6. Fascial closure instrument is introduced directly through anterior abdominal wall to help to maintain suture loop.
  7. The needle is removed, leaving the loop in place.
  8. The needle is entered again through the same skin puncture site around the medial half of the ring and enter the peritoneum, leaving a small space above the vas deferens and testicular vessels to avoid injury.
  9. The loop of suture is introduced into the hollow of the needle again and advance the suture into the first loop by the help of fascial closure.
  10. Withdraw the needle.
  11. Catch the suture end in the loop and withdraw them together then the suture is tied extra corporeally.

Patient outcomes:

Patients assessment and follow up:

1. Primary outcome measures:

   Operative time. Intraoperative complication. Rate of conversion to open surgery.
2. Secondary outcome measures:

1 and 3 months after the surgery to asses:

1. Cosmetic appearance: according to (The Scar Cosmesis Assessment and Rating "SCAR" Scale) [7].
2. Recurrence.
3. Hydrocele.
4. Testicular atrophy (postoperative imaging: > 50% loss of testicular volume or < 25% of volume of contralateral testis) [8].

ELIGIBILITY:
Inclusion Criteria:

* Include patients presented with inguinal hernia with age < 18 years.

Exclusion Criteria:

1. Age above 18 years.
2. Complicated inguinal hernia (e.g. irreducibility, obstruction and strangulation).
3. Pervious lower abdominal surgeries.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Operative time | during operation
  Operative time from start of incision making till end of operation and closure of incisions
Intraoperative complications | during operation
  as injury to inferior epigastric vessels, vas deferens and major pelvic vessels
Rate of conversion to open surgery. | during operation
  rate of conversion from laparoscopic surgery to open surgery.

SECONDARY OUTCOMES:
Cosmetic appearance | 1 and 3 months after the surgery
  according to (The Scar Cosmesis Assessment and Rating "SCAR" Scale)
Recurrence | 1 and 3 months after the surgery
  recurrence of inguinal hernia diagnosed clinically and/or by ultrasound
Hydrocele | 1 and 3 months after the surgery
  diagnosed clinically and/or by ultrasound
Testicular atrophy | 1 and 3 months after the surgery
  diagnosed clinically and/or by ultrasound (postoperative imaging: > 50% loss of testicular volume or < 25% of volume of contralateral testis).

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Cóbar, J. P., & Nichol, P. F. (2023). Introduction of pediatric laparoscopic inguinal hernia repair in Guatemala. BMC Surgery, 23(1). 2. Chang, S., Chen, J. Y., Hsu, C., Chuang, F., & Yang, S. S. D. (2015). The incidence of inguinal hernia and associated risk factors of incarceration in pediatric inguinal hernia: a nation-wide longitudinal population-based study. Hernia, 20(4), 559-563. 3. Elhosary, M. A., Elbatarny, A. M., Arafa, M., Mahmoud, S. M., Ismail, K. A., et al. (2023). Needlescopic primary paediatric inguinal hernia repair by hernia sac disconnection and peritoneal closure. Journal of Pakistan Medical Association, 73(4), S61-S66. 4. Maat, S. C., Dreuning, K. M. A., Nordkamp, S., Van Gemert, W., Twisk, J. W. R., et al. (2021). Comparison of intra- and extra-corporeal laparoscopic hernia repair in children: A systematic review and pooled data-analysis. Journal of Pediatric Surgery, 56(9), 1647-1656. 5. Hajong, R., Newme, K., & Moirangthem, T. (2022). A case control study of needlescopic herniotomy versus open herniotomy in children. Journal of Family Medicine and Primary Care, 11(7), 3633. 6. Shalaby, R., Negm, M., Elsawaf, M., Elsaied, A., Shehata, S., et al. (2021). Needlescopic disconnection and peritoneal closure for Pediatric inguinal hernia repair: a Novel technique. Surgical Laparoscopy Endoscopy & Percutaneous Techniques, 32(2), 272-278. 7. Kantor J, et al. Reliability and photographic equivalency of the SCAR Cosmesis assessment and rating (SCAR) scale, an outcome measure for postoperative scars. JAMA Dermatol. 2017;153(1):55-60 8. Ein, S.H. ∙ Nasr, A. ∙ Wales, P.W. ... Testicular atrophy after attempted pediatric orchidopexy for true undescended testis J Pediatr Surg. 2014; 49:317-322.